CLINICAL TRIAL: NCT04818970
Title: Adaptive Photo-Protection Trial: To Demonstrate the Safety and Efficacy of NB-UVB Light Therapy to Improve Outcomes in Hospitalized High-risk Patients With COVID-19
Brief Title: Photo-Protection Trial (NB-UVB vs. Placebo) in High-risk Hospitalized COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cytokind, Inc. (Industry)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other); Baylor College of Medicine (Other); West Jefferson Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPL0001-02
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Covid19; Corona Virus Infection; Autoimmune Diseases; Coagulation Disorder, Blood
Keywords: Narrow Band Ultraviolet Light B-Band; NB-UVB; Immune Dysregulation; Vitamin D
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Autoimmune Diseases; Blood Coagulation Disorders | interventions — Phototherapy

STUDY DESIGN:
Intervention Model Description: 1:1 Randomized Placebo Control Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Phototherapy of narrow band ultraviolet Light B-Band NB-UVB (Experimental): Daavlin Series 1 Phototherapy Unit that emits UVB light between 280nm and 320nm.
  Interventions: Device: Narrow Band ultraviolet B-Band Light
- Placebo - Light (Placebo Comparator): Daavlin Series 1 Phototherapy Unit that does not emit UVB light between 280nm and 320 nm.
  Interventions: Device: non Narrow Band ultraviolet B-Band Light

INTERVENTIONS:
Device: Narrow Band ultraviolet B-Band Light — Daily doses of NB-UVB for 8 consecutive days.
  Other Names: Phototherapy
  Arms: Phototherapy of narrow band ultraviolet Light B-Band NB-UVB
Device: non Narrow Band ultraviolet B-Band Light — Daily doses of non-NB-UVB for 8 consecutive days.
  Other Names: Placebo
  Arms: Placebo - Light

SUMMARY:
The purpose of this study to evaluate the translational application of the safe and effective treatment of Narrow-Band Ultraviolet light B-band (NB-UVB) to high-risk COVID-19 patients in an effort to improve their immune and hemostatic imbalance to increase survival and improve outcomes.

DETAILED DESCRIPTION:
Study Design

This is a multi-center, double blind, randomized control trial designed to assess the safety and efficacy of daily NB-UVB light for patients presenting to site hospitals over the age of 50 with a positive COVID-19 panel and at least one comorbidity.

This trial provides adjunctive therapy and no in-hospital treatments need to be modified in any way. The sponsor and the centers acknowledge standards of care are actively evolving and this trial is not intended to interfere in any form.

Double Blind: Patient and Health care provider will be blinded to the treatment vs. placebo by use of a non-NB-UVB light card. All dosing and times for treatment and placebo will be calculated the same methods.

Arm A: Control: Will receive non-NB-UVB light during the Treatment Period.

Arm B: Treatment: Will receive NB-UVB light during the Treatment Period.

Treatment Phase (Days 1-8): Treatment Schedule will be identical for arm A and B.

Follow Up Phase (Days 9-28 or discharge): Follow-up will be identical for arms A and B.

Blood Draw Schedule: Blood draws are to be performed after enrollment, before the first treatment day 1 and on days 3, 5, 8, 14 and day of discharge (if prior to day 14 unless blood draw has already occurred within one day of discharge).

ELIGIBILITY:
Inclusion Criteria:

-

To be eligible to enroll in the study, subjects must be:

* In-Hospital
* 50 years of age or older
* Hospitalized for COVID-I9 symptoms
* At least one comorbidity.
* They have taken a COVID-19 diagnostic test.
* Peripheral 02 saturation below 94 on room air, nasal cannula or non-rebreather
* Patients may remain enrolled as long as they remain hospitalized for
* COVID-19 symptoms and receive a positive test panel for COVID-19
* during the treatment phase
* Be able to provide consent.

Exclusion Criteria:

-

To be eligible to enroll in the study, subjects must not:

* Require ventilatory support at the time of enrollment.
* Concurrent pulmonary bacterial infection
* Taking Light Sensitive Medications
* Have Lupus Diagnosis
* Enrolled in an existing Covid-19 Trial
* Taking In-patient Vitamin oral Supplementation
* Severe mental or medical disability
* History of melanoma or dysplastic nevus syndrome
* Prisoner
* Active tuberculosis or Cystic Fibrosis, Severe Chronic Obstructive Pulmonary Disease (COPD) or Pulmonary Fibrosis requiring home supplemental oxygen
* Pre-existing pulmonary hypertension
* INR > 2, LFT 6 times greater than baseline
* Stage 3b CKD or ESRD diagnosis before COVID-19 onset
* Evidence of cirrhosis
* Evidence of pre-existing vascular disorder or coagulopathy
* Irreversible bleeding disorder
* Patients who are not full code
* Taking oral light sensitizing medications (See Appendix) or using light sensitizing topical
* medication in the phototherapy treatment zones
* Taking in patient or at home Vitamin D supplementation
* Have any photosensitive skin disorder such as Systemic Lupus Erythematosus, Porphyria or
* Pseudoporphyria, Polymorphous Light Eruption Xeroderma Pigmentosa, Chronic actinic
* dermatitis, Hydroa vacciniforme, Dermatomyositis Bloom Syndrome, Rothmund Thomas
* syndrome, Cockayne Syndrome
* Requiring oxygen supplementation via CPAP/BiPAP, ventilator support, High Flow Nasal
* Prong therapy (HFNP)
* Concurrent pulmonary bacterial infection at the time of enrollment
* Previous hospital admission for COVID-19 symptoms

Ages: 50 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Mortality Rate | 14 days
  % Patient Mortality
Mortality Rate | 28 days
  % Patient Mortality
WHO Ordinal Scale for Clinical Improvement | 14 days
  Improvement in WHO Ordinal Scale
WHO Ordinal Scale for Clinical Improvement | 28 days
  Improvement in WHO Ordinal Scale
Length of Hospital Stay | 28 days
  Days from Treatment to Discharge
Rate of Escalation to the ICU | day 14
  % of Patients Escalating to the ICU
Rate of Ventilator Support (intubation) requirement | day 28
  % of Patients Requiring Ventilator Support (intubation)

SECONDARY OUTCOMES:
Rate of Improved Immune Regulation as measured by (Any 3 of These): | 28 days
  1. Increased ratio of CD8 perforin to Monocyte IL6,
  2. Increased ratio ofNK perforin to Monocyte IL6
  3. Increased ratio of CD4 lFNg to Monocyte IL6
  4. Increased ratio of CD8 perforin to Monocyte TNF
  5. Increased ratio ofNK perforin to Monocyte TNF, and
  6. Increased ratio of CD4 IFNg to Monocyte TNF
Rate of Stabilization of the Immune Dysregulation (all 3 of These) | 28 days
  1. Decreased Th l and Th 17;
  2. Increased Th2;
  3. Increased circulating regulatory T Cells
Average Reduction in Inflammatory Markers: | 28 days
  HS-CRP (mg/L)
Average Reduction in Inflammatory Markers: | 28 days
  LDH (units per liter (U/L))
Average Reduction in Inflammatory Markers: | 28 days
  Ferritin (micrograms/L)
Improved Hemostatic Regulation by D-dimer Reduction | 28 days
  D-dimer (ng/mL)
Improved Hemostatic Regulation by reduce PTT | 28 days
  Partial Thromboplastin Time (PTT) Test
Average Reduced Viral Load. | 28 days
  Reduced viral load (copies/mL)
Average and Categorical Increase in Vitamin D: | 28 days
  1. 25(OH)D hydroxyvitamin D
     1. % of Patients Improving from Critical Deficiency (min. of 20ng/ml); ii. % of Patients Improving from Insufficiency (at min. of 30ng/ml);
  2. Active 1,25-dihydroxyvitamin D and
  i. % of Patients with Improvement from Insufficient (at min. of 18pg/ml);
% of Patients with a Change in oxygen requirement | 28 days
  1. Non-invasive positive pressure support (BiPAP & CPAP)
  2. Discharge from the ICU
  3. Removal from Ventilator Support
Average Temperature | 28 days
  1. (Average for each day) - Hospital Staff
  2. (Highest Record of the day) - Hospital Staff
Average Length of Hospitalization | 28 days
  Days in the ICU Days to Discharge Need for Rehospitalization Need for COVID Related Rehospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Frank H Lau, MD, Principal Investigator — Louisiana State University Health Sciences Center in New Orleans
Locations (1):
- West Jefferson Medical Center and LSUHSC-NO, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lau FH, Powell CE, Adonecchi G, Danos DM, DiNardo AR, Chugden RJ, Wolf P, Castilla CF. Pilot phase results of a prospective, randomized controlled trial of narrowband ultraviolet B phototherapy in hospitalized COVID-19 patients. Exp Dermatol. 2022 Jul;31(7):1109-1115. doi: 10.1111/exd.14617. Epub 2022 Jun 13. PMID 35638295